CLINICAL TRIAL: NCT02974907
Title: A Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of RGN-259 Ophthalmic Solutions for the Treatment of Dry Eye : ARISE-2
Brief Title: Assessment of the Safety and Efficacy of RGN-259 Ophthalmic Solutions for Dry Eye Syndrome : ARISE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ReGenTree, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-259/16-110-0008
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; Dry Eye; DES
MeSH Terms: conditions — Dry Eye Syndromes | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RGN-259 (Experimental): RGN-259: It is a preservative-free, sterile eye drop solution containing Tβ4
  Interventions: Drug: RGN-259
- Placebo (Placebo Comparator): It is composed of the same excipients as RGN-259 but does not contain Tβ4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGN-259 — A preservative-free, sterile eye drop solution containing Tβ4 for direct instillation into each eye, four times a day (QID) for 28 days
  Other Names: Tβ4; Thymosin Beta 4
  Arms: RGN-259
Drug: Placebo — It is composed of the same excipients as RGN-259 but does not contain Tβ4
  Other Names: Vehicle Control
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the safety and efficacy of RGN-259 Ophthalmic Solutions to placebo for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
Dry eye can be caused by many variable factors. Some examples include hormonal changes due to aging, or living in an environment of low humidity for long periods of time. Dry eye is a complex disease that may result in symptoms like discomfort, visual disturbance, and dryness. Patients with dry eye often have damage on the surface of the eye. In previous studies, RGN-259 has been shown to promote healing of the surface of the eye and decrease inflammation. It suggests that RGN-259 has a significant potential to be an important new safe and effective therapeutic in the treatment of dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye for at least 6 months
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months

Exclusion Criteria:

* Have any clinically significant slit-lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have ab uncontrolled systemic disease:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Ora Clinical Research and Development
Locations (1):
- Andover, MA, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened during a 14-day study run-in period prior to randomization. And after run-in period and confirmation of inclusion and exclusion criteria, all eligible subjects were randomized in a 1:1 ratio to receive 0.1% RGN-259 or placebo ophthalmic solution bilaterally, four times per day (QID) for 28 days. The study comprised of 5 visits over the course of approximately 6 weeks.
Groups:
- RGN-259: Active (0.1% RGN-259 ophthalmic solution)
- Placebo: Placebo (Placebo ophthalmic solution)
Period: Overall Study
Arm/Group | RGN-259 | Placebo
Started | 299 | 302
Completed | 286 | 292
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RGN-259 | Placebo | Total
Number analyzed (Participants) | 299 | 302 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.97) | 63.0 (11.48) | 62.5 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 223 | 438
  Male | 84 | 79 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 24 | 47
  Not Hispanic or Latino | 275 | 278 | 553
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 36 | 41 | 77
  White | 251 | 246 | 497
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Ocular Discomfort
Description: Change from Baseline at Day 29 using the Ora Calibra® Ocular Discomfort Scale (6-point scale where 0 = none and 5 = worst)
Time Frame: 29 days after first dosing
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 299 | 302
score on a scale | 0.07 [-0.05 to 0.19] | -0.04 [-0.15 to 0.08]

2. Primary Outcome: Corneal Fluorescein Staining
Description: Change from Baseline at Day 29 using the Ora Calibra® scale (5-point scale with half (0.5) increments where 0 = none and 4 = severe)
Time Frame: 29 days after first dosing
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 111 | 107
score on a scale | 0.07 [-0.06 to 0.20] | -0.01 [-0.13 to 0.12]

3. Secondary Outcome: Corneal Fluorescein Staining
Description: Comparing each of active group & Placebo.
Time Frame: 8, 15, 29 days after first dosing
Reporting Status: Not Posted

4. Secondary Outcome: Unanesthetized Schirmer's Test
Description: Comparing each of active group & Placebo.
Time Frame: 29 days after first dosing
Reporting Status: Not Posted

5. Secondary Outcome: Ocular Surface Disease Index (OSDI)©
Description: Comparing each of active group & Placebo.
Time Frame: 8, 15, 29 days after first dosing
Reporting Status: Not Posted

6. Secondary Outcome: Tear Film Break-Up Time
Description: Comparing each of active group & Placebo.
Time Frame: 8, 15, 29 days after first dosing
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Visual Acuity
Description: Change or shifts from Baseline
Time Frame: 1, 8, 15, 29 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Biomicroscopy Using the Slit-lamp
Description: Change or shifts from Baseline
Time Frame: 1, 8, 15, 29 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Adverse Event Query
Description: Frequencies
Time Frame: 1, 8, 15, 29 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Biomicroscopy Using the Undilated Fundoscopy
Description: Change or shifts from Baseline
Time Frame: 1, 29 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at every visit through study completion, up to Day 29.
Description: There was no anticipated/unanticipated deaths due to any cause in this study.
Arm/Group | RGN-259 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/302
Serious Adverse Events (participants affected / at risk) | 3/299 | 2/302
Other Adverse Events (participants affected / at risk) | 19/299 | 21/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGN-259 (N=299) | Placebo (N=302)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGN-259 (N=299) | Placebo (N=302)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 10 (12)
Eye Pain (Eye disorders) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (9) | 6 (6)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT02974907/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02974907/SAP_001.pdf